CLINICAL TRIAL: NCT01535976
Title: The Effect of Ketamine in The Prevention of Hypoventilation in Patients With and Without a Positive Berlin Questionnaire Undergoing Deep Sedation
Brief Title: Ketamine Infusion and Hypoventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Gildasio De Oliveira, M.D. Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STU00048723
Record Dates: First submitted 2011-09-09; First posted 2012-02-20 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-02

CONDITIONS: Hypoventilation
MeSH Terms: conditions — Hypoventilation | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): .9 normal saline infusion
  Interventions: Drug: Placebo
- Ketamine (Active Comparator): Infusion of ketamine
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Placebo — Placebo Comparator: Placebo
  .9 normal saline infusion
  Arms: Placebo
Drug: Ketamine — Ketamine infusion .5mg/kg bolus followed by 1.5 mcg/kg/minute until end of case
  Arms: Ketamine

SUMMARY:
Procedures performed under sedation have the same severity in regards to morbidity and mortality as procedures performed under general anesthesia1. The demand for anesthesia care outside the operating room has increased tremendously and it poses, according to a closed claim analysis, major risks to patients . Both closed claim analysis identified respiratory depression due to oversedation as the main risk to patients undergoing procedures under sedation. The major problem is that hypoventilation is only detected at very late stages in patients receiving supplemental oxygen. Besides the respiratory effects of hypoventilation, hypercapnia can also lead to hypertension, tachycardia, cardiac arrhythmias and seizures.

The incidence of anesthetized patients with obstructive sleep apnea has increased substantially over the last years along with the current national obesity epidemic. These patients are at increased risk of hypoventilation when exposed to anesthetic drugs. The context of the massive increase in procedural sedation and the extremely high prevalence of obstructive sleep apnea poses major respiratory risks to patients and it may, in a near future, increase malpractice claims to anesthesiologists. The development of safer anesthesia regimen for sedation are, therefore, needed. The establishment of safer anesthetics regimen for sedation is in direct relationship with the anesthesia patient safety foundation priorities. It addresses peri-anesthetic safety problems for healthy patient's. It can also be broadly applicable and easily implemented into daily clinical care.

Ketamine has an established effect on analgesia but the effects of ketamine on ventilation have not been clearly defined. The lack of validated and sensitive instruments to evaluate the effects of ketamine on ventilation is an important reason for the conflicting results.The investigators have demonstrated that the transcutaneous carbon dioxide monitor is accurate in detecting hypoventilation in patients undergoing deep sedation. Animal data suggest that when added to propofol in a sedation regimen, ketamine decreased hypoventilation when compared to propofol alone. It is unknown if ketamine added to a commonly used sedative agent (propofol) can decrease the incidence and severity of hypoventilation in patients undergoing deep sedation. It is also unknown if the effect of ketamine on ventilation are different in patients with and without obstructive sleep apnea.

The investigators hypothesized that patients receiving ketamine and propofol will develop less intraoperative hypoventilation than patients receiving propofol alone. The investigators also hypothesized that this effect will be even greater in patients with obstructive sleep apnea than patients without obstructive sleep apnea.

Significance: Respiratory depression due to oversedation was identified twice as the major factor responsible for claims related to anesthesia. The high prevalence of obstructive sleep apnea combined with more complex procedures done in outpatient settings can increase physical risks to patients and liability cases to anesthesiologists. The main goal of this project is to establish the effect of ketamine in preventing respiratory depression to patients undergoing procedures under sedation. If the investigators confirm the their hypothesis , their findings can be valuable not only to anesthesiologist but also to other specialties ( Emergency medicine, gastroenterologists, cardiologists, radiologists) that frequently performed procedural sedation. The research questions is;does ketamine prevent hypoventilation during deep sedation? The hypotheses is; ketamine will prevent hypoventilation during sedation cases.

ELIGIBILITY:
Inclusion Criteria:

* ASA I,II
* Age 18-64
* Females undergoing surgical procedures requiring sedation

Exclusion Criteria:

* Pregnant subjects
* Breastfeeding
* Patients or surgeon request

  ---Drop Out:
* Patient or surgeon request,
* Conversion to general anesthesia
* Inability to obtain data from Co2 monitor

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio De Oliveira, MD, Principal Investigator — Northwestern University
Locations (1):
- Prentice Womens Hospital, Chicago, Illinois, United States

REFERENCES:
- [Derived] De Oliveira GS Jr, Fitzgerald PC, Hansen N, Ahmad S, McCarthy RJ. The effect of ketamine on hypoventilation during deep sedation with midazolam and propofol: a randomised, double-blind, placebo-controlled trial. Eur J Anaesthesiol. 2014 Dec;31(12):654-62. doi: 10.1097/EJA.0000000000000025. PMID 24247410

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospital based recruitment. From August 2011 to June 2012.
Groups:
- Ketamine: Infusion of ketamine
  Ketamine : Ketamine infusion .5mg/kg bolus followed by 1.5 mcg/kg/minute until end of case
- Placebo: .9 normal saline infusion
  Placebo : Placebo Comparator: Placebo
  .9 normal saline infusion
Period: Overall Study
Arm/Group | Ketamine | Placebo
Started | 27 | 27
Completed | 26 | 26
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ketamine: Infusion of ketamine
  Ketamine : Ketamine infusion .5mg/kg bolus followed by 1.5 mcg/kg/minute until end of case along with propofol 100 mcg/kg/min
- Placebo: normal saline infusion
  Placebo : Placebo Comparator: Placebo
  normal saline infusion along with propofol 100 mcg/kg/min
- Total: Total of all reporting groups
Arm/Group | Ketamine | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (7.67) | 46.89 (7.35) | 47.65 (7.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Hypoventilation
Description: Subjects receiving intraoperative ketamine in addition to propofol will demonstrate less hypoventilation during the surgical procedure.
Time Frame: 8 hours
Population: The median percentage of the sedation time with TCO2 > 50 mmHg
Measure: Median (95% Confidence Interval); unit: % time
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 26 | 26
% time | 1.2 (95) [0 to 83] | 65 [0 to 88]

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Ketamine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

LIMITATIONS AND CAVEATS:
We did not use depth of anesthesia monitor guided protocol due to controversial effects of ketamine of the correlation of processed EEG monitor and clinical levels of sedation. We did not use opioids as part of the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No